CLINICAL TRIAL: NCT00244426
Title: II Italian Study on Atrial Fibrillation (S.I.F.A. II): Prevention of Thromboembolic Events in Patients With Non Valvular Atrial Fibrillation.
Brief Title: S.I.F.A. II: Prevention Of Thromboembolic Events In Patients With Nonrheumatic Atrial Fibrillation
Acronym: SIFA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 293-CVD-9010-004; A7651004
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
Keywords: Prevention of thromboembolic events in patients with non valvular atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — indobufen; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: indobufen
- 2 (Active Comparator)
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: indobufen — Indobufen capsules 100 and 200mg
  Arms: 1
Drug: aspirin — Acetylsalicylic acid capsules 300mg
  Arms: 2

SUMMARY:
Evaluate efficacy and safety of Indobufen v. Aspirin in preventing thromboembolic events in patients at high risk of CV events such as patients suffering from nonrheumatic atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or paroxysmal non rheumatic atrial fibrillation with cardioembolic risk factors: hypertension, ischemic cardiopathy, Congestive Heart Failure, diabetes mellitus

Exclusion Criteria:

* Clinically relevant organ disease
* creatinine clearance < 30 ml/min
* gastric or duodenal ulcer
* severe anaemia or poliglobulia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2000-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
combined endpoints: cerebral ictus (ischemic or haemorragic), cardiovascular death, nonfatal acute myocardial infarction (AMI) or peripheral embolism. The first event occurring during the study will be considered. | 3.5 years

SECONDARY OUTCOMES:
Global mortality, ischemic ictus, disabling ictus, TIA, nonfatal acute myocardial infarction, fatal and nonfatal hemorrhagic events, fatal and nonfatal embolisms. | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- Italy (115):
  - Pfizer Investigational Site, Lagosanto, FE
  - Pfizer Investigational Site, Perugia, PG
  - Pfizer Investigational Site, Poggibonsi, SI
  - Pfizer Investigational Site, Siena, SI
  - Pfizer Investigational Site, Busto Arsizio, VA
  - Pfizer Investigational Site, Peschiera del Garda, VR
  - Pfizer Investigational Site, Abbadia S. Salvatore (SI)
  - Pfizer Investigational Site, Acquaviva Delle Fonti (BA)
  - Pfizer Investigational Site, Albano Laziale
  - Pfizer Investigational Site, Alessandria
  - Pfizer Investigational Site, Ancona
  - Pfizer Investigational Site, Angera
  - Pfizer Investigational Site, Antella
  - Pfizer Investigational Site, Aosta
  - Pfizer Investigational Site, Arezzo
  - Pfizer Investigational Site, Assisi
  - Pfizer Investigational Site, Asti
  - Pfizer Investigational Site, Avellino
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Bentivoglio
  - Pfizer Investigational Site, Bergamo
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Brindisi
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Carbonia
  - Pfizer Investigational Site, Casarano
  - Pfizer Investigational Site, Casarano (LE)
  - Pfizer Investigational Site, Caserta
  - Pfizer Investigational Site, Cassano Delle Murge (BA)
  - Pfizer Investigational Site, Castelfranco Veneto
  - Pfizer Investigational Site, Castiglion Del Lago
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Catanzaro
  - Pfizer Investigational Site, Cesena
  - Pfizer Investigational Site, Chieti
  - Pfizer Investigational Site, Cirie (TO)
  - Pfizer Investigational Site, Citta' Di Castello (Pg)
  - Pfizer Investigational Site, Cittadella
  - Pfizer Investigational Site, Città della Pieve
  - Pfizer Investigational Site, Copertino
  - Pfizer Investigational Site, Cosenza
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Desio
  - Pfizer Investigational Site, Eboli (SA)
  - Pfizer Investigational Site, Faenza
  - Pfizer Investigational Site, Fidenza
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Foligno
  - Pfizer Investigational Site, Forlimpopoli (Fo)
  - Pfizer Investigational Site, Forlì
  - Pfizer Investigational Site, Frosinone
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Giulianova
  - Pfizer Investigational Site, Gorizia
  - Pfizer Investigational Site, Gracciano (Si)
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Gubbio
  - Pfizer Investigational Site, Gubbio (PG)
  - Pfizer Investigational Site, Imperia
  - Pfizer Investigational Site, Latina
  - Pfizer Investigational Site, Lecce
  - Pfizer Investigational Site, Livorno
  - Pfizer Investigational Site, Lucca
  - Pfizer Investigational Site, L’Aquila
  - Pfizer Investigational Site, Macerata
  - Pfizer Investigational Site, Mantova
  - Pfizer Investigational Site, Martina Franca
  - Pfizer Investigational Site, Matera
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Mestre
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Moncalieri to
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Orvieto Scalo
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pescara
  - Pfizer Investigational Site, Piombino
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Pistoia
  - Pfizer Investigational Site, Popoli (Pe)
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Pozzilli
  - Pfizer Investigational Site, Prato
  - Pfizer Investigational Site, Ravenna
  - Pfizer Investigational Site, Reggio Emilia
  - Pfizer Investigational Site, Rho (MI)
  - Pfizer Investigational Site, Rimini
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, S. Giovanni Rotondo
  - Pfizer Investigational Site, San Bonifacio
  - Pfizer Investigational Site, San Felice A Cancello
  - Pfizer Investigational Site, San Giovanni Rotondo
  - Pfizer Investigational Site, San Vito al Tagliamento
  - Pfizer Investigational Site, Sant' Omero ( Te)
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Savigliano
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Taranto
  - Pfizer Investigational Site, Telese Terme
  - Pfizer Investigational Site, Termoli
  - Pfizer Investigational Site, Todi
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Torre Del Greco (NA)
  - Pfizer Investigational Site, Trieste
  - Pfizer Investigational Site, Udine
  - Pfizer Investigational Site, Varese
  - Pfizer Investigational Site, Velletri
  - Pfizer Investigational Site, Vibo Valentia
  - Pfizer Investigational Site, Vicenza
  - Pfizer Investigational Site, Vigevano
  - Pfizer Investigational Site, Viterbo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=293-CVD-9010-004&StudyName=S.I.F.A.%20II%3A%20Prevention%20Of%20Thromboembolic%20Events%20In%20Patients%20With%20Nonrheumatic%20Atrial%20Fibrillation.